CLINICAL TRIAL: NCT05084131
Title: Feasibility of Online Visit Format for Post-Operative Visit After Colon and Rectal Surgery
Brief Title: Web-based Visit for Colorectal Surgery
Acronym: Web-visit
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Justin Maykel, Division Chief of Colorectal Surgery, University of Massachusetts, Worcester
Other Study IDs: H00017264
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Surgery
Keywords: online visit; web visit; patient portal; colorectal surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Use of an online questionnaire as follow-up after abdominal colorectal surgery — Patients were asked to complete a questionnaire via the institutional patient portal. Participants were also asked to upload a photo of their respective incisions. Participants then had an in-person follow-up visit.

SUMMARY:
The purpose of this study to evaluate how well an online format would work for the first post-operative visit after a patient undergoes colon and rectal surgery. This online format is integrated into Epic MyChart. This study aims to determine whether the online format is feasible and acceptable to patients and surgeons as a standard post-operative visit.

DETAILED DESCRIPTION:
Participants were asked to complete a post-operative survey using an online patient portal, EPIC MyChart, after elective abdominal colon or rectal resection. Participants were also asked to do upload a picture of their incisions. Colorectal surgeons reviewed responses/pictures and communicated concerns/recommendations via the same patient portal. At the in-person follow-up visit, both patients and colorectal surgeons completed a satisfaction survey regarding the both visit types.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Planned/underwent surgery that was performed by a surgeon in the Division of Colon and Rectal Surgery
3. Requires a post-operative follow-up outpatient visit 2-3 weeks from surgery or from discharge from hospital
4. Has access to a smart mobile phone, tablet or computer to access online web interface for the web-based visit
5. Patients with an Epic MyChart account set up.
6. Has ability to take photographs of surgical incision or has access to someone who can take a picture for them.

Exclusion Criteria:

1. Requires visiting nurse services at discharge from hospital
2. Cannot use web-based interface or unable to complete questions online
3. Cannot read English, speak English, or would require interpreter services. The reason for excluding these patients is there are not yet MyChart services available in non-English languages at Umass Memorial. It would not be fiscally possible to acquire these for a pilot feasibility study. As the MyChart experience is meant to be completed at home, it would not be possible to provider a medical interpreter in a non-office or hospital setting.
4. Adults unable to consent (adults lacking capacity)
5. Individuals who are not yet adults (infants, children, teenagers)
6. Prisoners
7. Pregnant women
8. Patients undergoing anal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent elective abdominal colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with questionnaire | 2 weeks
  After the in-person follow-up visit, patients were asked to complete a satisfaction questionnaire of the online visit survey
Provider satisfaction with questionnaire | 2 weeks
  After the in-person follow-up visit, colorectal surgeons were asked to complete a satisfaction survey

CONTACTS AND LOCATIONS:
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beauharnais CC, Hill SS, Sturrock PR, Davids JS, Alavi K, Maykel JA. Efficacy and satisfaction of asynchronous TeleHealth care compared to in-person visits following colorectal surgical resection. Surg Endosc. 2022 Dec;36(12):9106-9112. doi: 10.1007/s00464-022-09383-8. Epub 2022 Jun 17. PMID 35713720